CLINICAL TRIAL: NCT02264093
Title: Effects on the Airway Lumen of Single Oral Doses of Talsaclidine (12, 24, 48 and 60 mg) in Combination With a Single Oral Doses of 160 mg Propranolol in Comparison to the Effects of the Monosubstances (60 mg Talsaclidine and 160 mg Propranolol) in Healthy Elderly Male Volunteers (Partially Randomised, Open Label, Intraindividual Comparison)
Brief Title: Effects on the Airway Lumen of Talsaclidine in Combination With Propranolol in Comparison to the Effects of the Monosubstances in Healthy Elderly Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 506.114
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Propranolol; talsaclidine fumarate

ARMS (3):
- Talsaclidine with Propranol (Experimental)
  Interventions: Drug: Propranolol; Drug: Talsaclidine
- Propranolol (Active Comparator)
  Interventions: Drug: Propranolol
- Talsaclidine (Active Comparator)
  Interventions: Drug: Talsaclidine

INTERVENTIONS:
Drug: Propranolol
  Arms: Propranolol; Talsaclidine with Propranol
Drug: Talsaclidine
  Arms: Talsaclidine; Talsaclidine with Propranol

SUMMARY:
To investigate the effects on airway lumen of talsaclidine in combination with propranolol and of talsaclidine and propranolol given as monosubstances

ELIGIBILITY:
Inclusion Criteria:

All participants in the study should be healthy males, range from 50 to 65 years of age and be within +- 20% of their normal weight (Broca-Index).

Exclusion Criteria:

* Volunteers will be excluded from the study if the result of the medical examination or laboratory tests (especially those which indicate liver malfunction) are judged by the clinical investigator to differ significantly from the normal clinical values
* Volunteers with blood pressure lower than 120/80 mm Hg or pulse rate below 60 beats/min
* Volunteers whose blood pressure dropped below 100/60 mm Hg in the pre-test within 80 mg propranolol
* Volunteers with Raw-values higher than their predicted normal upper limit
* Volunteers with known gastrointestinal, hepatic , renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with disease of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with known history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with history of allergy / hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Volunteers who have taken a drug with a long half life (>=24 hours) within at least one month or less than ten half lives of the respective drug before enrolment in the study
* Volunteers who received any other drugs which might influence the results of the trial during the week prior the start of the study
* Volunteers who have participated in another study with an investigational drug within the last 2 month preceding this study
* Volunteers who are unable to refrain from smoking on the study days
* Volunteers who smoke more than 10 cigarettes (or 3 cigars or pipes) per day
* Volunteers who drink more than 40 g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who have donated blood (>=100ml) within the last 4 weeks
* Volunteers who participated in excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1999-11; Primary Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Airway resistance (Raw) | Up to 8 hours after drug administration
Specific conductance (SGaw) | Up to 8 hours after drug administration
Forced expiratory volume in 1 sec (FEV1) | Up to 8 hours after drug administration

SECONDARY OUTCOMES:
Number of participants with clinically significant findings in vital signs | Up to 8 days after last drug administration
Number of participants with clinically significant findings in laboratory tests | Up to 8 days after last drug administration
Number of participants with adverse events | Up to 8 days after last drug administration
Cmax (maximum measured concentration of the analyte in plasma) | Up to 12 hours after drug administration
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | Up to 12 hours after drug administration
AUC (area under the plasma concentration versus time curve) | Up to 12 hours after drug administration